CLINICAL TRIAL: NCT00826813
Title: Phase IV Study of Self-Expandable Esophageal Stent Loaded With 125I Seeds: a Randomized Controlled Multiple Center Trial in Patients With Advanced Esophageal Cancer
Brief Title: Trial Using 125I Embedded Stent in Patients With Advanced Esophageal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Southeast University, China (Other)
Responsible Party: Xiao-Hui Chen, MD, Zhongda Hospital, Department of Radiology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009A123456; H200343
Record Dates: First submitted 2009-01-21; First posted 2009-01-22 (Estimated); Last update posted 2009-01-22 (Estimated); Status verified 2009-01

CONDITIONS: Esophageal Cancer
Keywords: Dysphagia; esophageal cancer; stent; brachytherapy
MeSH Terms: conditions — Esophageal Neoplasms; Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- stenting (Experimental): The conventional esophageal stent or 125I radiation stent is placed in the patients with dysphagia who are enrolled to the study.
  Interventions: Device: Esophageal stent placement

INTERVENTIONS:
Device: Esophageal stent placement — The esophageal stent combined a self-expandable covered esophageal stent and 125I radioactive seeds. Sheathes were attached to the outer surface of the stent, containing 125I radioactive seeds of CIAE 6711. The seeds were loaded into the sheathes on the stent immediately before implantation of the stent. The numbers and dose of the radioactive stent seeds was determined by the treatment plan system based on the size of the individual tumor. To cover the entire lesion of the tumor by the sheaths containing 125I seeds, at least 2 cm exceeding the tumor margins was required. The distance between the two sheaths was 15mm. In the control group, conventional covered esophageal stents were used which provided by the same company as those attached with 125I seeds.
  Other Names: esophageal stent implantation

SUMMARY:
More than half of patients with esophageal cancer are inoperable because of late stage cancer or metastasis and they have to undergo palliative treatments. Dysphagia is the major symptom of patients with inoperable esophageal cancer. To relieve the dysphagia and improve the quality of life of such patients, stent placement has been widely accepted to be an option for palliation of the symptoms. However, recurrence of the neoplastic stricture remains a challenge after stent placement. To combine the advantages of the immediate relief of the esophageal dysphagia with the stent placement and radiation therapy with brachytherapy, a novel esophageal stent loaded with 125I seeds has been developed in the authors' institute. The preliminary clinical trial in a single institute has demonstrated better results than the conventional stent. This prospective multiple center trial is designed to further demonstrate the clinical outcomes with this irradiation, stent in patients compared to those using a conventional covered stent.

DETAILED DESCRIPTION:
Esophageal cancer ranks as the fourth leading cause of death from cancer in China and sixth worldwide. Although the prognosis of surgical resection for esophageal cancer has been improved, more than 50% of such patients are inoperable and have to undergo palliative treatments because of late stage cancer or metastasis. Dysphagia is the predominate symptom of patients with inoperable esophageal cancer. To relieve the dysphagia and improve the quality of life of such patients, brachytherapy has previously been utilized. Recently, stent placement has been widely accepted to be an option for palliation of the symptoms due to the esophageal strictures. However, recurrence of the neoplastic stricture remains a challenge after stent placement. To combine the advantages of the immediate relief of the esophageal dysphagia with the stent placement and radiation therapy with brachytherapy, a novel esophageal stent loaded with 125I seeds has been developed in the authors' institute. The technical feasibility and safety with this new stent has been demonstrated to be adequate in a healthy rabbit model. The following preliminary clinical study in a single institute has demonstrated longer survival time, better quality of life and less restenosis of the stent than whose with the conventional stent. This prospective multiple center trial is designed to further demonstrate the clinical outcomes with this irradiation, stent in patients compared to those using a conventional covered stent.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary cancer of esophagus,
* Must be dysphagia caused by esophageal cancer,
* Without esophageal fistulas,
* Must be an inpatient,
* Life expectancy is over 6 months

Exclusion Criteria:

* Esophageal fistulas,
* Tracheal compression with symptoms,
* WBC <2000/mm3 and Platelet count <50,000/mm3,
* Concurrent therapies after stenting:surgery, chemotherapy,radiotherapy, Traditional Chinese Medicine

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2009-01; Primary Completion 2010-03 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Death of the patient

SECONDARY OUTCOMES:
Quality of life | 3, 6, 12 months
Restenosis of the stent | 3, 6, 12 months
Dysphagia relief | 3, 6, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gao-Jun Teng, MD, Ph.D, Principal Investigator — Zhongda Hospital
Locations (1):
- #87 Dingjiaqiao Road, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Guo JH, Teng GJ, Zhu GY, He SC, Fang W, Deng G, Li GZ. Self-expandable esophageal stent loaded with 125I seeds: initial experience in patients with advanced esophageal cancer. Radiology. 2008 May;247(2):574-81. doi: 10.1148/radiol.2472070999. Epub 2008 Mar 18. PMID 18349316
- [Background] Guo JH, Teng GJ, Zhu GY, He SC, Deng G, He J. Self-expandable stent loaded with 125I seeds: feasibility and safety in a rabbit model. Eur J Radiol. 2007 Feb;61(2):356-61. doi: 10.1016/j.ejrad.2006.10.003. Epub 2006 Nov 7. PMID 17085003